CLINICAL TRIAL: NCT02864849
Title: Total Neoadjuvant Induction and Consolidation CapeOX Plus Neoadjuvant Intensity Modulated Radiotherapy With Concurrent Capecitabine for MRI Defined High-risk Rectal Cancer
Brief Title: Total Neoadjuvant Induction and Consolidation CapeOX Plus IMRT With Capecitabine for MRI Defined High-risk Rectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Aiwen Wu, Chief, Unit III & Ostomy Service, Gastrointestinal Cancer Center, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUCH-R02
Record Dates: First submitted 2016-08-04; First posted 2016-08-12 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; neoadjuvant; radiotherapy; chemotherapy; toxicity
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Capecitabine; Radiotherapy, Intensity-Modulated

ARMS (1):
- TNT (Experimental): Patients with MRI defined high-risk rectal cancer will receive chemotherapy before and after chemoradiation, and will not receive adjuvant treatment. This arm is called total neoadjuvant treatment (TNT). The neoadjuvant chemotherapy regimen is designed as 3 cycles of CapeOX (Capecitabine+Oxaliplatin) over a period of approximately 8 weeks. Tumor response will be evaluated after chemotherapy. Then patients will undergo 22f-IMRT (Intensity modulated radiotherapy) with capecitabine. Patients will receive two more cycles of consolidation CapeOX if tolerable when there was no progressed disease in induction CapeOX.
  Finally, patients will receive TME (Total mesorectal excision) following TNT if no metastasis occurs.
  Interventions: Drug: Oxaliplatin; Drug: Capecitabine; Radiation: Intensity modulated radiotherapy; Procedure: Total mesorectal excision

INTERVENTIONS:
Drug: Oxaliplatin
  Other Names: OXA
Drug: Capecitabine
  Other Names: CAPE
Radiation: Intensity modulated radiotherapy
  Other Names: IMRT
Procedure: Total mesorectal excision
  Other Names: TME

SUMMARY:
This study is designed to test the efficacy and safety of total neoadjuvant induction and consolidation CapeOX plus neoadjuvant intensity modulated radiotherapy with concurrent capecitabine for MRI defined high-risk rectal cancer.

DETAILED DESCRIPTION:
This phase II trial is studying the efficacy and safety of total neoadjuvant treatment for MRI defined high-risk locally advanced rectal cancer.

MRI imaging features as mrT3c/T3d/T4a/T4b, threatening circumferential resection margin, mrN2 disease or extramural vascular invasion are defined as high-risk factor and proved to associated with unfavorable oncological outcome, especially for distant metastasis. Induction and consolidation chemotherapy plus radiation may increase both systemic and local control. Total neoadjuvant treatment schedule also has advantages as improved patient tolerance, early closure of defunctioning ileostomy etc.

In this study, patients with MRI defined high-risk rectal cancer will receive 3 cycles induction CapeOX, intensity modulated radiotherapy with concurrent capecitabine and 2 cycles consolidation CapeOX and Total mesorectal excision.

The induction chemotherapy related G3-4 toxicity occurred in 42% of patients in GCR-3 trial (23% during RT, 19% during induction chemotherapy). It is hypothesized that the neoadjuvant chemotherapy related G3-4 toxicity rate of the present regimen will be lower than 25% (10% during IMRT, 15% during induction/consolidation chemotherapy). A sample size of 67 achieves 80% power to detect a difference (△P =17%, P1=25%, P0=42%) using a one-sided binomial test. (α= 0.05). If the number of G3-4 toxic event is 21 or less, the hypothesis that P1>= 42% is rejected. About 10 % loss to follow-up was anticipated, so an additional eight patients will be recruited. The study requires 75 subjects in all.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤75 years.
* ECOG Performance status 0-1.
* Histologically confirmed diagnosis of adenocarcinoma of the rectum.
* The distance from down verge of tumor to anal-rectal junction (ARJ) ≤8cm based on MRI, or ≤12 cm based on sigmoidoscopy.
* Clinical Stage T3c, T3d, T4a or T4b, or EMVI (+) or mrN2 or CRM (+) based on MRI.
* No evidence of distant metastases.
* No prior pelvic radiation therapy.
* No prior chemotherapy or surgery for rectal cancer.
* No active infections requiring systemic antibiotic treatment.
* ANC > 1.5 cells/mm3, HGB > 10.0 g/dL, PLT > 100,000/mm3, total bilirubin ≤ 1.5 x ULN, AST≤ 3 x ULN, ALT ≤ 3 x ULN.
* Patients must read, agree to, and sign a statement of Informed Consent prior to participation in this study.

Exclusion Criteria:

* Recurrent rectal cancer.
* Anticipated unresectable tumor after neoadjuvant treatment.
* Creatinine level greater than 1.5 times the upper limit of normal.
* Patients who have received prior pelvic radiotherapy.
* Patients who are unable to undergo an MRI.
* Patients with a history of a prior malignancy within the past 5 years, except for adequately treated basal cell or squamous cell skin cancer.
* Patients with a history of any arterial thrombotic event within the past 6 months. This includes angina (stable or unstable), MI, TIA, or CVA.
* Other Anticancer or Experimental Therapy.
* Women who are pregnant or breast-feeding.
* Patients with any other concurrent medical or psychiatric condition or disease which would make them inappropriate candidates for entry into this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2016-08; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Major adverse events | 3 years
  Adverse events will be graded using the NCI Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0

SECONDARY OUTCOMES:
Disease-free survival (DFS) | 3 years
  The 3-year DFS will be defined as the percentage of patients alive without local recurrence or distant metastasis of disease at 3 years measured from the date of the administration of treatment.
Pathological downstaging rate | 1 year
  The pathological result for each patient will be compared with MRI pre-stage and re-stage and downstaging rate will be recorded.
Compliance rate with neoadjuvant treatment schedule | 1 year
  To measure the compliance rate to the total neoadjuvant treatment schedule.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Core 30 (EORTC QLQ-C30) | Time0: before neoadjuvant treatment; Time1: at 4 months after the completion of neoadjuvant radiation; Time2: 12 months after Time1; Time3: 24 months after Time1; Time4: 36 months after Time1
  EORTC QLQ-C30 (Aaronson et al., 1993). The questionnaire assesses health status and quality of life of cancer patients using 30 items grouped in one global scale, five multi-item functioning scales, three symptom scales and six single symptom items.
  The items are scored on a four-point Likert scale with higher scores indicating a better level of functioning or a higher level of symptoms. The validity and reliability of the Mandarin versions of the questionnaire have been established.
European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Colorectal Cancer Module 29 (EORTC QLQ-CR29) | Time0: before neoadjuvant treatment; Time1: at 4 months after the completion of neoadjuvant radiation; Time2: 12 months after Time1; Time3: 24 months after Time1; Time4: 36 months after Time1
  EORTC QLQ-CR29 (Whistance et al., 2009). The questionnaire measures health-related quality of life in patients with colorectal cancer, using 29 items grouped in four functional scale and 18 symptom scale.
  The items are scored on a four-point Likert scale with higher scores indicating a better level of functioning or a higher level of symptoms. The validity and reliability of the Mandarin versions of the questionnaire have been established.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China